CLINICAL TRIAL: NCT07035080
Title: Efficacy Of Isokinetic Strength Training On Functional Performance In Children With Hemophilia
Brief Title: Isokinetic Strength Training On Functional Performance
Acronym: Isokinetic
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Sara Yousef Abdel Elglil Yousef Elsebahy, lecture of pediatric physical therapy, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KFSIRB200-497
Record Dates: First submitted 2025-06-09; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Hemophilia
MeSH Terms: conditions — Hemophilia A | interventions — Electric Stimulation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Experimental): the control group will receive traditional treatment program for one hour per session including (ultrasound stretching and strengthening exercise )
  Interventions: Other: tradional physical therapy
- group 2 (Experimental): the study group will receive interferential therapy in addition to the same treatment program given to the control groups.
  Interventions: Other: interferential therapy

INTERVENTIONS:
Other: interferential therapy — Thirty hemophilic males (type A and B) children with unilateral hemarthrosis, age ranged from 8 to 12 years participated in this study. They were selected from the outpatient clinic. Faculty of physical therapy, kafrelsheik university. The patients were divided randomly into two groups of equal number , control and study groups, 15 patients each . the control group (7 left and 8 right hemarthrosis) received traditional treatment program for one hour per session includeing (ultrasound stretching and strengthening exercise ) , while the study group (6 left and 9 right hemarthrosis) received interferential therapy in addition to the same treatment program given to the control groups.
  Arms: group 2
Other: tradional physical therapy — Thirty hemophilic males (type A and B) children with unilateral hemarthrosis, age ranged from 8 to 12 years participated in this study. They were selected from the outpatient clinic. Faculty of physical therapy, kafrelsheik university. The patients were divided randomly into two groups of equal number , control and study groups, 15 patients each . the control group (7 left and 8 right hemarthrosis) received traditional treatment program for one hour per session includeing (ultrasound stretching and strengthening exercise ) , while the study group (6 left and 9 right hemarthrosis) received interferential therapy in addition to the same treatment program given to the control groups.
  Arms: group 1

SUMMARY:
Hemophilia is a congenital , recessive clotting disease featured by cerebra ( The most dangerous ) and musculoskeletal (the most common and disabling) hemorrhages . It is a gender -specific coagulopathy resulting from a factor VIII (F VIII) deficiency in hemophilia A and factor IX (F IX) deficiency in hemophilia B( Felip et al., 2011) Loss of muscle mass is typical of hemophilia arthropathy, There are two basic reasons that account for such muscle loss. The first reason is due to inactive joints as the result of long -term immobilization that hemophilic patients are obliged to do because of continuous lesions in muscles and joints, and the second reason is a decrease in physical exercise by hemophilic patients because of the risk of lesions that they face (Toca-Herrera et al., 2008).

Interferential therapy is a type of transcutaneous electrical nerve stimulation (TENS). Two slightly different, medium frequency- alternating currents are simultaneously applied to the affected area through electrodes. Superpisition or interference between the currents causes the combined electrical current to rise and fall (Burch et al, 2008).

Low amplitude modulated frequencies elicit a "beating" or "tapping" sensation and muscle twitch response, while higher amplitude modulated frequencies elicit "buzzing" or "tingling sensation" and titanic muscle contraction ( Defrin et al., 2007).

Several methods are available for testing muscle strength. These include manual muscle testing and dynamometry includes the use of handheld dynamometers, handgrip dynamometers, and isokinetic dynamometers (Sisto and Dyson-hudson, 2007).

Isokinetic dynamometers measure torque produced at the anatomic joint throughout the available range of motion (ROM). Isokinetic dynamometers. Such as the kinCom (Chatanooga Corp, Chatanooga, Tennessee). Biodex (Biodex Medical systems. Inc) and Lido Active isokinetic System (Loredan, Inc, Davis , California ) measure torque by controlling the velocity of the movement and measuring the force applied via a force transducer (Sisto and Dyson-hunson, 2007).

Isokinetic test record the torque produced throughout the entire ROM and allow for the identification of regions of strength or weakness within the range ( Remauld et al., 2005).

Isokinetic assessment has primarily been recommended for strength testing as maximal force is applied during all phase of the movement at a constant velocity . The isokinetic mode is also safe to use with children because there is minimal risk of the muscle and joint injuries that can results from efforts to control the load if using free weights in one repetition -maximum testing (Mark et al., 2003).

DETAILED DESCRIPTION:
Loss of muscle mass is typical of hemophilia arthropathy, There are two basic reasons that account for such muscle loss. The first reason is due to inactive joints as the result of long -term immobilization that hemophilic patients are obliged to do because of continuous lesions in muscles and joints, and the second reason is a decrease in physical exercise by hemophilic patients because of the risk of lesions that they face (Toca-Herrera et al., 2008).

With time , hemophilic arthropahy results in weak and unstable joints. The patient is also very vulnerable to stressful locomotors stimulation, which, in turn, causes greater instability and risk of lesions. This cicious circle of pain immobility , atrophy , joint instability , and new hemorrhagic episodes may eventually lead to total invalidity ( Gomis et al., 2009).

ELIGIBILITY:
Inclusion Criteria:

* Patients of both groups (study and control groups ) were selected according to the following criteria:

  1. Each group contained 15 male children. They were suffering from unilateral knee heamarthrothesis .
  2. The joint problems (pain and bleeding ) ranges from mild to moderate according to the classification of hemophilia recommended by the Orthopedic advisory committee of the World Federation of hemophilia (appendix 1) (Holder and Cotta, 1989).
  3. Patients were able to stand and walk independently.
  4. They had no neurological or psychological problems.
  5. All patients were clinically and medically stable.
  6. They were able to understand the requirements of the study.
  7. They were suffering from moderate hemophilia.
  8. They were not suffering from acute joint and muscle bleeds during treatment time.
  9. None of the children suffered from fixed deformities of the affected lower limb.
  10. All the children received the same medical treatment to control bleeding.
  11. They had no visual no hearing deficits B. Exclusion criteria

  <!-- -->

  1. Patients with advanced radiographic changes including:

     * Bone destruction.
     * Bony ankylosis .
     * Knee joint subluxation.
     * Epiphyseal fracture.
  2. Patients who had congenital or acquired skeletal deformities in both lower limbs.
  3. Patients who had any neurological deficits such as convulsions involuntary movements or those receiving muscle relaxants.

     Exclusion Criteria:

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-06-20 (Estimated); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
changes in muscle strength | after 3 months

SECONDARY OUTCOMES:
change in level of pain | after 3 months
change in function ability | after 3 months

IPD SHARING:
Plan to Share IPD: Undecided